CLINICAL TRIAL: NCT05758116
Title: A Prospective, Open-label, Single-arm, Phase II Trial Investigating the Efficacy and Safety of Tislelizumab Consolidation Therapy After Radiotherapy or Sequential Chemoradiation in Locally Advanced NSCLC Patients
Brief Title: Tislelizumab Consolidation Therapy After Radiotherapy or Sequential Chemoradiation in Locally Advanced NSCLC Patients
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Peking University Cancer Hospital & Institute (Other)
Responsible Party: Principal Investigator, rongyu, Professor, Peking University Cancer Hospital & Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022YJZ46
Record Dates: First submitted 2023-02-17; First posted 2023-03-07 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-11

CONDITIONS: Non-small Cell Lung Cancer; Consolidation Immunotherapy; Radiotherapy or Sequential Chemoradiation
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — tislelizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Consolidation Tislelizumab (Experimental): Patients completed radiotherapy alone or sequential chemoradiation with 42 days received consolidation Tislelizumab 200mg every 3 weeks for 12 months.
  Interventions: Drug: Tislelizumab

INTERVENTIONS:
Drug: Tislelizumab — Tislelizumab: 200mg d1,q21d*17

SUMMARY:
The current standard of care for locally advanced non-small cell lung cancer (NSCLC) is concurrent chemoradiation and consolidation immunotherapy. In real world clinical practice, patients who cannot tolerate concurrent chemoradiation generally received radiotherapy alone or sequential chemoradiation. These patients are more likely to develop distant metastases and therefore may require tolerable systemic consolidation regimens. However, there is a lack of evidence from clinical studies on consolidation immunotherapy after radiotherapy alone or sequential chemoradiation. The aim of the study is to explore the efficacy and safety of Tislelizumab consolidation therapy after radiotherapy or sequential chemoradiation in locally advanced NSCLC patients who are intolerable of concurrent concurrent chemoradiation.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with stage III(AJCC 8th) unresectable NSCLC, or resectable but intolerant or refusing surgery;
2. Intolerable of concurrent chemoradiation;
3. No progression after radiotherapy or sequential chemoradiation;
4. Chemotherapy: standard dose of 2-6 cycles of paclitaxel, pemetrexed or gemcitabine in combination with platinum; Radiotherapy: starting within 3 months after chemotherapy using IMRT or VMAT technique. The target volume includes the primary tumor and regional lymph nodes, and the prescription dose 95% PTV ranges from 50Gy to 66Gy;
5. ECOG PS0-2;
6. PD-L1≥1%;
7. Age≥18 years, and life expectancy>3 months;
8. Adequate Hematologic, biochemistry and organ function (to be confirmed by test results within 7 days prior to the first dose);
9. Be able to provide written informed consent (ICF) and able to understand and agree to comply with study requirements and assessment schedule.

Exclusion Criteria:

1. Patients with EGFR-sensitive mutations and ALK rearrangements;
2. Any prior use of anti-PD-1, anti-PD-L1, or anti-cytotoxic T-lymphocyte-associated antigen-4 (CTLA-4) antibodies (including Ipilimumab or any other antibody targeting the T-cell co-stimulation or checkpoint pathway);
3. History of allergy to components of Tislelizumab;
4. Any active malignancy within 2 years prior to enrollment, except for the specific cancers examined in this study and any locally recurrent cancers that have been eradicated (e.g., resected basal or squamous cell skin cancer, superficial bladder cancer, cervical or breast cancer in situ);
5. History of interstitial lung disease or pneumonia requiring oral or intravenous steroids;
6. Progression after radiotherapy or sequential chemoradiation;
7. Unresolved ≥grade2 toxicities from radiotherapy and sequential chemoradiation, (excluding those that the investigator determines do not affect study treatment, such as alopecia);
8. Grade 2 or severe Pneumonia from radiotherapy or sequential chemoradiation;
9. Administration of a live vaccine within 30 days prior to treatment start (seasonal influenza vaccine without live vaccine is allowed);
10. Severe chronic or active infections (including tuberculosis infections, etc.) requiring systemic antibacterial, antifungal or antiviral therapy ≤ 14 days prior to treatment start;
11. History of immunodeficiency, including a positive HIV test, or other acquired or congenital immunodeficiency disease, or a history of organ transplantation;
12. History of active autoimmune disease requiring systemic therapy;
13. Treatment with long-term systemic immunosuppressive medications (≥10 mg/d prednisone or equivalent doses of other steroids) or other immunosuppressive medications;
14. History of uncontrolled cardiovascular disease; or clinically significant QT interval prolongation, or QTc interval >480 ms during screening period;
15. Abnormal liver function [total bilirubin > 1.5 times of the upper limit of normal value; ALT/AST > 2.5 times of the upper limit of normal value in patients without liver metastases and ALT/AST > 5 times of the upper limit of normal value in patients with liver metastases], abnormal renal function (serum creatinine > 1.5 times of the upper limit of normal value);
16. History of serious concomitant diseases (e.g., severe hypertension, diabetes, thyroid disease, active infection, etc.) ;
17. History of diagnosed neurological or psychiatric disorders, including epilepsy or dementia;
18. Unsuitable for participation in this study assessed by investigators;
19. Patients who were already enrolled in other clinical studies;
20. Mixed lung cancer with small cell components.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-07-07 (Actual); Primary Completion 2025-07-07 (Estimated); Study Completion 2026-07-07 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | 6 months after enrollment
  Defined from the date of enrollment to the date of death or any recurrence.

SECONDARY OUTCOMES:
Overall survival | From date of enrollment to maximum of 3 years or death
  Defined from the date of enrollment to the date of death.
Objective response rate | From date of enrollment to maximum of 3 years or death
  Defined as the occurrence of a complete or partial response per RECIST 1.1 criteria.
Treatment-related adverse events | Duration of treatment and follow up until death or 3 years after enrollment
  Graded according to NCI-CTCAE v5.0

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University Cancer Hospital and Institute, Beijing, China

IPD SHARING:
Plan to Share IPD: No